CLINICAL TRIAL: NCT02323776
Title: Correlation of Radiotherapy-related Features With Postoperative Complications in Patients With Esophageal Cancer Treated With Trimodality Therapy
Brief Title: Defining the Radiotherapy Dose and Volume Parameters Affecting Postoperative Complications in Esophageal Cancer Patients
Status: Terminated | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 14-28-03/09
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Trimodality protocol — neoadjuvant chemoradiotherapy followed by surgery

SUMMARY:
The purpose of this study is to identify features of the cumulative dose-volume histogram (DVH) for patients treated with trimodality therapy in oesophageal cancer and correlate these with postoperative complications.

DETAILED DESCRIPTION:
Intention to treat analysis in patients initially assigned to be treated with the trimodality protocol: neoadjuvant chemoradiotherapy followed by surgery.

The investigators will retrospectively evaluate several parameters of the treatment planning of patients treated with a preoperative regimen (CROSS regimen 41,4 Gy in 23 fractions or 50, 4 Gy in 28 fractions ):

* PTV volume1
* MLD, V30, V20, V15, V10, VS5 (Volume lung less dan 5 Gy)2 (lung toxicity)
* MHD, V20, V30, V403 (heart toxicity)
* Mean stomach dose, V50 stomach
* Mitochondrial DNA if available per patient Pre-existing cardiac,pulmonary comorbidity, smoking behavior, BMI, type of surgery and chemotherapy (especially taxanes) will be scored and take into account in a multivariate analysis. The investigators will collect these data and correlate the data with the presence of postoperative complications, time of onset of complications and duration of hospitalization. These latter data are already scored in a prospective manner at the Atrium Medical Center in Heerlen.

ELIGIBILITY:
Inclusion Criteria:

* Oesophageal cancer patients
* initially treated with a preoperative dose of radiation in combination with chemotherapy and subsequently undergone surgical resection

Exclusion Criteria:

* Patients who were treated with definitive chemoradiation or palliative radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Oesophageal cancer patients who were initially treated with a preoperative dose of radiation in combination with chemotherapy and who subsequently underwent surgical resection at the Atrium Hospital in Heerlen. All patients were included in a prospectively maintained database.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | within 30 and 90 Days after operation
  Cardiac complications (arrhythmia etc )
  * Respiratory complications (pneumonia, pleural effusion etc)
  * Anastomotic leakage
  * Postoperative 30-day mortality
  * Total postoperative mortality
  * Treatment-related mortality
  * Hospitalization and stay at intensive care unit duration

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Netherlands